CLINICAL TRIAL: NCT01283035
Title: A Phase II Study of MK-2206 in the Treatment of Recurrent High-Grade Serous Platinum-Resistant Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: A Phase II Study of Akt Inhibitor MK2206 in the Treatment of Recurrent Platinum-Resistant Ovarian, Fallopian Tube, or Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00549; NCI-2013-00549 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10-402 (Other: Dana-Farber Cancer Institute); 8729 (Other: CTEP); P30CA006516 (NIH)
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Results first posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-05

CONDITIONS: Ovarian Sarcoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — MK 2206

ARMS (1):
- Treatment (Akt inhibitor MK2206) (Experimental): Akt inhibitor MK2206 will be taken PO once a week for four weeks (one cycle). Treatment will continue for as long as a subject is benefiting from the study drug.
  Interventions: Drug: Akt Inhibitor MK2206; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Akt Inhibitor MK2206 — Given PO
  Other Names: MK2206
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
Akt inhibitor MK2206 is a drug that may stop cancer cells from growing by blocking a protein called protein kinase B (AKT) inside the cell. AKT interacts with other proteins in the cell that are part of the P13K/AKT pathway, a pathway that is know to play a role in the growth of cancer cells. Mutations in P13K or in AKT, or changes in another protein called phosphatase and tensin homolog (PTEN) in this pathway can lead it to become more active than is normal. This study investigates how effective MK-2206 is in treating ovarian, fallopian tube, or primary peritoneal cancer where there are mutations in P13K or AKT or low levels of PTEN.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the activity of MK-2206 (Akt inhibitor MK2206) in patients with recurrent grade 2 or 3 platinum-resistant high-grade serous ovarian, fallopian tube, or peritoneal cancer, as measured by the frequency of patients experiencing an objective tumor response by Response Evaluation Criteria In Solid Tumors (RECIST) criteria or who survive progression-free for at least 6 months after initiation of therapy.

SECONDARY OBJECTIVES:

I. To assess the duration of progression-free and overall survival following initiation of therapy with MK-2206 in the cohort of patients enrolled on this study.

II. To determine the toxicities of MK-2206, as assessed by the active version of the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0 III. To explore the association between select biomarkers and response to MK-2206 (as assessed by objective tumor response, progression-free survival, and overall survival) IV. To explore the development of feedback loop activation and target inhibition with MK-2206 via analysis of pre-treatment and post-treatment biopsies in select patients enrolled in the trial.

OUTLINE:

Akt inhibitor MK2206 will be taken orally (PO) once a week for four weeks (one cycle). Treatment will continue for as long as a subject is benefiting from the study drug.

During each cycle subjects will have a physical exam, blood samples and an electrocardiogram (EKG) (first 2 cycles). Every 2 cycles a computed tomography (CT) scan or magnetic resonance imaging (MRI) of chest, stomach area, and pelvis will be performed. Optional tumor biopsies may be performed.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed high grade (grade 2 or 3) serous ovarian, fallopian tube, or primary peritoneal cancer; participants with mixed histology are eligible if the serous component is the dominant histological subtype
* Participants must have measurable disease as defined by RECIST 1.1 criteria
* Participants must have evidence of a defect in the PI3K/AKT pathway, defined by A) evidence of loss of PTEN by immunohistochemistry in a CLIA-certified assay or B) documentation of PIK3CA or AKT mutation in a CLIA-certified assay; for patients without prior CLIA-certified evidence of a PI3K/AKT pathway defect, PTEN testing will be performed by immunohistochemistry in a CLIA-certified assay; availability of a formalin fixed paraffin embedded (FFPE) block of cancer tissue from the original or most recent biopsy must be available for mutational and immunohistochemical analysis
* Prior therapy:

  * Prior chemotherapy must have included a first-line platinum-based regimen with or without consolidation chemotherapy
  * Patients may have received up to 2 lines of therapy (including cytotoxic or biological and/or targeted therapies) in the recurrent setting
  * Prior hormonal therapy is acceptable and will not count as an additional line of therapy
  * Patients may not have previously received prior AKT or PI3 kinase pathway inhibitors (including mTOR inhibitors)
  * Patients should have platinum-resistant disease, where platinum resistance is defined as having progressive disease within 6 months of receipt of prior platinum therapy
* Life expectancy of greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Karnofsky > 60%)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 8.0 g/dL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) < 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits or creatinine clearance > 60 mL/min/1.73 m^2 for subjects with creatinine levels about institutional normal
* Toxicities of prior therapy (excepting alopecia) should be resolved to less than or equal to grade 1 as per NCI-CTCAE v4.0
* Patients must be able to tolerate oral medications and not have gastrointestinal illnesses that would preclude absorption of MK-2206
* The effects of MK-2206 on the developing human fetus are unknown; for this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study
* Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered to grade 1 or less (excepting alopecia) due to agents administered more than 4 weeks earlier
* Participants may not be receiving any other study agents
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-2206
* Participants receiving any medications or substances that are strong inhibitors or inducers of CYP450 3A4 are ineligible; lists including medications and substances known or with the potential to interact with the CYP450 3A4 isoenzymes are provided in Appendix C; if the participant is taking any agent known to affect or with the potential to affect CYP450 3A4 isoenzymes, this should be discussed with the overall PI
* Preclinical studies demonstrated the potential of MK-2206 for induction of hyperglycemia in all preclinical species tested; patients with diabetes or at risk for hyperglycemia are eligible for this study, but the hyperglycemia should be well controlled on oral agents before the patient enters the trial; a fasting serum glucose of > 130 mg/dL or a HgbA1c > 7.5 mg/dL will exclude patients from entry on study; patients requiring insulin for control of their hyperglycemia are excluded from entry on this study
* Preclinical studies indicated transient changes in QTc interval during MK-2206 treatment; prolongation of QTc interval is potentially a safety concern while on MK-2206 therapy; cardiovascular: baseline QTcF > 450 msec (male) or QTcF > 470 msec (female) will exclude patients from entry on study; a list of medications that may cause QTc interval prolongation are listed in Appendix D, and should be avoided by patients entering on trial
* Due to a high incidence of bradycardia by Holter monitor, preexisting significant heart block or baseline bradycardia due to cardiac disease will exclude patients from treatment with MK-2206
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Current signs and/or symptoms of bowel obstruction
* Current dependency on IV hydration or TPN
* Pregnant women are excluded from this study because MK-2206 is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with MK-2206, breastfeeding should be discontinued if the mother is treated with MK-2206; these potential risks may also apply to other agents used in this study
* Individuals with a history of a different malignancy are ineligible except for the following circumstances; individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy; individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: breast cancer in situ, cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin
* Human immunodeficiency virus (HIV)-positive individuals on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with MK-2206; iIn addition, these individuals are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated
* Patients may not use natural herbal products or other "folk remedies" while participating in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Liu, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Akt Inhibitor MK2206)
Started | 6
Completed | 5
Not Completed | 1
Not completed — Subject later found ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Efficacy (as Measured by Objective Response Rate) of Akt Inhibitor MK2206 in Patients With Recurrent High-grade Platinum-resistant Serous Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Description: If 4 or more of the final set of 29 patients demonstrate a response, then the null hypothesis H0: =< 5% can be rejected in favor of the alternative hypothesis H1: >= 20% with an alpha of 0.05 and beta of 0.20 (i.e., 80% power).
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progression, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression
Time Frame: Up to 3 years
Population: Five patients started study treatment.
Measure: Number; unit: participants
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 5
participants
  Stable Disease | 4
  Progressive Disease | 1

2. Secondary Outcome: Association Between Select Biomarkers and Response to Akt Inhibitor MK2206 (as Assessed by Objective Tumor Response, Progression-free Survival, and Overall Survival)
Description: The frequency of mutations in the PI3K/AKT and RAS pathways, copy number alterations, and PTEN loss and AKT expression as assessed by IHC will be tabulated. Associations between these markers with clinical outcome such as response rate and duration of PFS will be assessed.
Time Frame: Up to 3 years
Population: Minimal activity was observed and patient accrual was slow. This analysis was not completed as the data was not collected.
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 0

3. Secondary Outcome: Development of Feedback Loop Activation and Target Inhibition With Akt Inhibitor MK2206 Via Analysis of Pre-treatment and Post-treatment Biopsies in Select Patients Enrolled in the Trial
Time Frame: Up to 3 years
Population: as for outcome 2
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Overall Survival Following Initiation of Therapy With Akt Inhibitor MK2206 in the Cohort of Patients Enrolled on This Study
Description: Distributions will be estimated using Kaplan-Meier analysis.
Time Frame: Up to 3 years
Population: as for outcome 2
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 0

5. Secondary Outcome: Duration of Progression-free Following Initiation of Therapy With Akt Inhibitor MK2206 in the Cohort of Patients Enrolled on This Study
Description: Distributions will be estimated using Kaplan-Meier analysis.
Time Frame: Up to 3 years
Population: as for outcome 2
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 0

6. Secondary Outcome: Toxicities of Akt Inhibitor MK2206, as Assessed by the Active Version of the NCI Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Time Frame: Up to 3 years
Population: Number of participants experiencing toxicities.
Measure: Number; unit: participants
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 5
participants | 5

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the initiation of the study intervention, throughout the study, and within 30 days of the last study intervention.
Arm/Group | Treatment (Akt Inhibitor MK2206)
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Akt Inhibitor MK2206) (N=5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)
Colonic Obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Akt Inhibitor MK2206) (N=5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Chelitis (Gastrointestinal disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Increased urea (Investigations) | 1 (1)
Oral mucositis (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Throat tightening (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less